CLINICAL TRIAL: NCT00605982
Title: Breast MRI as a Preoperative Tool for DCIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-124
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Ductal Carcinoma in Situ
Keywords: MRI
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

ARMS (1):
- 1 (Experimental): Women with core biopsy proven DCIS with or without microinvasion seen for surgical consultation at Memorial Sloan-Kettering Cancer Center and for whom operative intervention is planned.
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — The patient will then undergo a breast MRI as part of their preoperative work-up of DCIS. Biopsy of any suspicious areas by needle biopsy or at the time of surgery. If appropriate, repeat MRI after biopsy or surgery. Follow-up for 10 years (you will be contacted once a year to see how you are doing).

SUMMARY:
Breast MRI is a fairly new technology, but it has been well studied. It is now used routinely in many patients with breast cancer. It has been shown to be useful in detecting areas of cancer that cannot be seen using other types of scans or tests.

The purpose of this study is to see how often MRI can find other areas of cancer in women with one area of breast cancer, and to determine how having the MRI test affects their treatment. The purpose is also to study any areas of abnormality seen on your MRI with special methods that allow the images of your breast tissue and the microscopic analysis of your breast tissue to be compared very carefully. The study also aims to follow women who enter the study over a 10-year period to determine how often the breast cancer comes back.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 60 at time of consent
* Clinical stage is consistent with Stage 0 or Stage I T1mic at presentation
* Core biopsy proven DCIS or DCIS with microinvasion (invasion ≤0.1 cm), prior to enrollment
* Breast surgery to be performed at MSKCC
* Informed consent obtained
* Female

Exclusion Criteria:

* Age 60 or over at time of consent
* Patients who are pregnant or nursing
* Patients with contraindications to breast conservation
* Excisional biopsy of DCIS or DCIS with microinvasion, prior to enrollment
* Patients with any contraindications to MRI including pacemaker, tissue expander, other metallic surgical implants, weight over 350 lb., previous gadolinium reaction, metal fragments in eye

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2006-10-10 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
To prospectively evaluate the value of preoperative breast MRI in women with core biopsy-proven DCIS. | conclusion of the study

SECONDARY OUTCOMES:
To determine the proportion of all patients in this study in whom breast MRI identifies at least one site of cancer separate from the index lesion. | conclusion of the study
To estimate re-excision rates and mastectomy rates in patients with DCIS undergoing preoperative MRI. | conclusion of the study
To estimate the proportion of patients with DCIS in which preoperative MRI will change surgical planning. | conclusion of the study
To estimate the long-term ipsilateral breast recurrence rate in women with DCIS undergoing preoperative breast MRI. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Van Zee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org